CLINICAL TRIAL: NCT05130203
Title: Developing and Assessing an Innovative Exergaming Technology for Older Adults Living in Long-term Care Homes With a User-centered Design Approach
Brief Title: Developing and Assessing an Innovative Exergaming Technology for Older Adults Living in Long-term Care Homes
Acronym: MouvMat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Charlene Chu, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00693
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Physical Inactivity; Cognitive Decline; Aging; Social Isolation
Keywords: nursing homes; long-term care; exergaming; user-centered design; older adult; aging; depression; dementia
MeSH Terms: conditions — Sedentary Behavior; Cognitive Dysfunction; Social Isolation; Depression; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MouvMat Exergaming (Experimental): Older adults in the intervention group will participate in a 6-week, 3 times per week, 45 minutes per session exercise program involving use of the MouvMat. Each resident from the intervention group will engage with the exergame supervised by a qualified and trained RA. Each intervention session will involve groups of 4-5 participants, with participants taking turns. An RA blinded to participants' condition will collect the outcome data.
  Interventions: Behavioral: MouvMat Exergaming
- Standard Recreational Programming (Other): A control group will meet on a similar schedule as the MouvMat group for standard recreational programming conducted by onsite recreational therapists. The same RA from the experimental group will collect outcome measurements from control group participants.
  Interventions: Behavioral: Standard Recreational Programming

INTERVENTIONS:
Behavioral: MouvMat Exergaming — Sessions engaging with exergaming device.
  Arms: MouvMat Exergaming
Behavioral: Standard Recreational Programming — Conducted by recreational therapists.
  Arms: Standard Recreational Programming

SUMMARY:
Residents living in long-term care (LTC) homes spend up to 75% of their day in sedentary, socially withdrawn situations which increases their risk for depression, dementia, decreased functional status and increased care costs. Physical activity is an accepted intervention to improve the physical health, cognition, and well-being of older adults. Moreover, systematic reviews have found that exergaming (i.e. physical activity gamified with technology) offers physical, cognitive, and social benefits by means of dual-task activities that engage both motor and cognitive abilities. The effect of exergaming for older adults in LTC is less clear, as this population has greater health needs related to physical health conditions, cognitive impairment, and functional dependence. Given the increased global demand for LTC, there is a need to develop and assess innovative exergaming technologies that can support the physical and cognitive health of LTC residents.

MouvMat is an exergaming technology intervention with an interactive digital gaming surface designed for older adults (OA) in LTC settings. Participants can play familiar games, like Simon or Bingo, by stepping on or tapping the surface with an assistive pointing device. Games can be played individually or with multiple players. LED lights on the surface provide an adaptive digital display and embedded pressure sensors respond to players' input. The investigators collaboratively designed a preliminary prototype with OA aged 65 and older in a pilot project.

The overall objective of this proposal is to conduct a pilot RCT of the Mouvmat to evaluate the feasibility, acceptability and efficacy of the exergaming technology to improve the primary outcome of mobility, and the secondary outcomes of cognitive function and social isolation compared to a usual care control group receiving standard recreational programming by recreational therapists.

DETAILED DESCRIPTION:
The sample size calculation was completed based on an effect size of 0.65 (power = 0.80; 2-tailed; α= 0.05). Assuming a 5% attrition rate, a total of 56 residents (28 people in a control group and 28 people in the intervention group) will be recruited. A block randomization design using a number generator to conceal the randomization sequence will be used to assign participants' units to the intervention or control groups. Block randomization was conducted to comply with COVID-19 restrictions. The investigators will attempt to recruit equal numbers of men and women with a range of mobility requirements (i.e., ambulate independently, using gait aids such as canes or walkers). In addition, a mix of approximately 5-10 LTC staff and/or residents' family members will be recruited at the end of the trial to conduct semi-structured interviews to understand the acceptability of the technology, design, usability and enjoyment, potential facilitators and barriers to exergame technology.

ELIGIBILITY:
Inclusion Criteria:

* All residents at the participating long-term care homes are eligible if they are 55 years of age or older
* Ability to communicate and speak English
* Able to provide informed consent or have a substitute decision maker (SDM) who provides informed consent
* A family member, friend, or personally-hired caregiver of an older adult residing in one of our participating LTC facilities are eligible to participate if they are 18 years of age or older, can communicate and speak English
* The LTC resident does not need to be enrolled in or study in order for their family member/friend/caregiver to participate
* LTC staff are eligible if they can communicate and speak English, are currently working in one of the participating LTC facilities, have at least 6 months experience working with older adults in LTC, providing or supervising physical or recreational activities, or involved with purchasing or directing these activities, and are a member of one of the following professions/positions: physiotherapist, physiotherapy assistant, recreational therapist, or LTC administrator.

Exclusion Criteria:

* Residents will be ineligible to participate in the study is they cannot communicate or speak English
* Residents who typically do not participate in recreational activities
* Residents who have a severe sensory (e.g., deaf, blind) or severe to moderate cognitive impairment AND/OR scores less than 20 on the Mini- Mental Status Examination (MMSE)
* Family Members who cannot communicate or speak English
* Family Members who cannot interact with the MouvMat due to sensory limitations (i.e., severe visual or auditory impairment)
* Family Members who cannot provide verbal feedback

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean mobility scores on the Timed-up-and-Go test | Baseline and mid-point of the intervention (3 weeks)
  Completion time in seconds when participant sits in a standard armchair and is instructed to stand up and walk to a line 3 m away at their normal pace, turn around and sit back down in the chair.
Change in mean mobility scores on the Timed-up-and-Go test | Baseline and following the completion of the intervention (6 weeks)
  Completion time in seconds when participant sits in a standard armchair and is instructed to stand up and walk to a line 3 m away at their normal pace, turn around and sit back down in the chair.
Change in mean mobility scores on the 2-Minute Walk Test | Baseline and mid-point of the intervention (3 weeks)
  Distance walked in meters when a participant is instructed to walk at the fastest speed that they can for 2 minutes.
Change in mean mobility scores on the 2-Minute Walk Test | Baseline and following the completion of the intervention (6 weeks)
  Distance walked in meters when a participant is instructed to walk at the fastest speed that they can for 2 minutes.
Adverse events (e.g. injury) related to exergame use | Over the course of the intervention (baseline to 6 weeks)
  Number of adverse events related to use of the exergame in the intervention group
Feasibility related to adherence rate | Over the course of the intervention (baseline to 6 weeks)
  Mean percentage of sessions attended in the intervention group (i.e., number of sessions attended / total scheduled sessions)

SECONDARY OUTCOMES:
Change in mean working memory scores on digit span | Baseline and mid-point of the intervention (3 weeks)
  Total scores for the WAIS-III forward and backward digit span, in which participants are asked to repeat a series of digits that are read by an experimenter in the same order (forward) or reverse order (backward).
Change in mean working memory scores on digit span | Baseline and following the completion of the intervention (6 weeks)
  Total scores for the WAIS-III forward and backward digit span, in which participants are asked to repeat a series of digits that are read by an experimenter in the same order (forward) or reverse order (backward).
Change in mean basic attention/psychomotor speed on the Trail Making Test A | Baseline and mid-point of the intervention (3 weeks)
  Time to completion in seconds on a task requiring connecting numbered dots on a page in order as quickly as possible.
Change in mean basic attention/psychomotor speed on the Trail Making Test A | Baseline and following the completion of the intervention (6 weeks)
  Time to completion in seconds on a task requiring connecting numbered dots on a page in order as quickly as possible.
Change in mean alternating attention scores on the Trail Making Test B | Baseline and mid-point of the intervention (3 weeks)
  Time to completion in seconds on a task requiring switching between connecting numbers and letters in dots on a page as quickly as possible.
Change in mean alternating attention scores on the Trail Making Test B | Baseline and following the completion of the intervention (6 weeks)
  Time to completion in seconds on a task requiring switching between connecting numbers and letters in dots on a page as quickly as possible.
Change in errors made on an alternating sequences test | Baseline and mid-point of the intervention (3 weeks)
  Number of errors made on a task requiring alternating between drawing two designs. This test is sensitive to cognitive problems with executive functions including inhibition and perseveration.
Change in errors made on an alternating sequences test | Baseline and following the completion of the intervention (6 weeks)
  Number of errors made on a task requiring alternating between drawing two designs. This test is sensitive to cognitive problems with executive functions including inhibition and perseveration.
Change in mean verbal fluency scores | Baseline and mid-point of the intervention (3 weeks)
  Number of words generated in one minute given a letter cue
Change in mean verbal fluency scores | Baseline and following the completion of the intervention (6 weeks)
  Number of words generated in one minute given a letter cue
Change in mean scores for social isolation assessed by UCLA Loneliness Scale 3 | Baseline and mid-point of the intervention (3 weeks)
  Total score on a 20-item questionnaire that assesses how often a person feels lonely and isolated from others.
Change in mean scores for social isolation assessed by UCLA Loneliness Scale 3 | Baseline and following the completion of the intervention (6 weeks)
  Total score on a 20-item questionnaire that assesses how often a person feels lonely and isolated from others.
Change in mean scores on the Cornell Scale for Depression in Dementia | Baseline and mid-point of the intervention (3 weeks)
  Total scores on a measure based on interviews on 19 items related to depression.
Change in mean scores on the Cornell Scale for Depression in Dementia | Baseline and following the completion of the intervention (6 weeks)
  Total scores on a measure based on interviews on 19 items related to depression.

OTHER OUTCOMES:
Acceptability on a version of the modified Treatment Evaluation Inventory (m-TEI) adapted for exergame use | Following the completion of the intervention (6 weeks)
  Mean total score from intervention group participants and family members/staff
Semi-structured interviews to evaluate the acceptability of the technology, design, usability and enjoyment, potential facilitators and barriers | Following the completion of the intervention (6 weeks)
  A semi-structured interview will be completed with residents in the intervention group, as well as stakeholders including family members and staff, with questions designed to understand the acceptability of the technology, design, usability and enjoyment, potential facilitators and barriers to exergame technology. The post-intervention interviews will be analyzed using thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Charlene Chu, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Chester Village, Toronto
  - Kensington Gardens, Toronto

REFERENCES:
- [Background] Ikezoe T, Asakawa Y, Shima H, Kishibuchi K, Ichihashi N. Daytime physical activity patterns and physical fitness in institutionalized elderly women: an exploratory study. Arch Gerontol Geriatr. 2013 Sep-Oct;57(2):221-5. doi: 10.1016/j.archger.2013.04.004. Epub 2013 May 9. PMID 23664785
- [Background] Chu CH, Puts M, Brooks D, Parry M, McGilton KS. A Feasibility Study of a Multifaceted Walking Intervention to Maintain the Functional Mobility, Activities of Daily Living, and Quality of Life of Nursing Home Residents With Dementia. Rehabil Nurs. 2020 Jul/Aug;45(4):204-217. doi: 10.1097/rnj.0000000000000186. PMID 30325875
- [Background] Shankar A, McMunn A, Demakakos P, Hamer M, Steptoe A. Social isolation and loneliness: Prospective associations with functional status in older adults. Health Psychol. 2017 Feb;36(2):179-187. doi: 10.1037/hea0000437. Epub 2016 Oct 27. PMID 27786518
- [Background] de Souto Barreto P, Morley JE, Chodzko-Zajko W, H Pitkala K, Weening-Djiksterhuis E, Rodriguez-Manas L, Barbagallo M, Rosendahl E, Sinclair A, Landi F, Izquierdo M, Vellas B, Rolland Y; International Association of Gerontology and Geriatrics - Global Aging Research Network (IAGG-GARN) and the IAGG European Region Clinical Section. Recommendations on Physical Activity and Exercise for Older Adults Living in Long-Term Care Facilities: A Taskforce Report. J Am Med Dir Assoc. 2016 May 1;17(5):381-92. doi: 10.1016/j.jamda.2016.01.021. Epub 2016 Mar 21. PMID 27012368
- [Background] Beard JR, Officer A, de Carvalho IA, Sadana R, Pot AM, Michel JP, Lloyd-Sherlock P, Epping-Jordan JE, Peeters GMEEG, Mahanani WR, Thiyagarajan JA, Chatterji S. The World report on ageing and health: a policy framework for healthy ageing. Lancet. 2016 May 21;387(10033):2145-2154. doi: 10.1016/S0140-6736(15)00516-4. Epub 2015 Oct 29. PMID 26520231
- [Background] Chu CH, Biss RK, Cooper L, Quan AML, Matulis H. Exergaming Platform for Older Adults Residing in Long-Term Care Homes: User-Centered Design, Development, and Usability Study. JMIR Serious Games. 2021 Mar 9;9(1):e22370. doi: 10.2196/22370. PMID 33687337